CLINICAL TRIAL: NCT05465200
Title: Coordinated Treatment of Cardiogenic Shock Patients in Lower Silesia, Poland
Brief Title: Lower Silesia Cardiogenic Shock Initiative
Acronym: LSCSI
Status: Recruiting | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Wiktor Kuliczkowski, Head of Catheterization Laboratory, Wroclaw Medical University
Other Study IDs: WMU012021
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic shock; ECMO; Heart transplant; Mechanical circulatory support; Impella
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Structured treatment of cardiogenic shock patients — Creation of hub&spoke structure which covers all Lower Silesian Voivodeship (Poland) for treatment of cardiogenic shock patients. Based on shared protocol patients are reported to "hub" by "spoke" and decision is made as for patient transfer or further treatment in the "spoke" facility. If decision on transfer is made, patient is further treated according to "hub" on site shock team protocol

SUMMARY:
LSCSI is a Hub&Spoke project with the main aim to improve the outcome of patients with cardiogenic shock in Lower Silesia region, Poland. It consists of one "hub" which is Wroclaw University Hospital and eleven "spokes" which are eleven cardiology departments situated in Lower Silesian Voivodeship. The consortium have unified protocol defining which cardiogenic shock patient and when should be transferred to the "hub" for enhanced treatment options including durable mechanical circulatory support or heart transplant. The "hub" have 7/24 Shock Team on-site supplied with a protocol how to proceed with "spoke" transferred patients including decision making on which mechanical circulatory support implant with subsequent de-escalation or escalation pathway.

DETAILED DESCRIPTION:
LSCSI is a Hub&Spoke project with the main aim to improve the outcome of patients with cardiogenic shock in Lower Silesia region, Poland. It consists of one "hub" which is Wroclaw University Hospital and eleven "spokes" which are eleven cardiology departments situated in Lower Silesian Voivodeship. The consortium have unified protocol defining which cardiogenic shock patient and when should be transferred to the "hub" for enhanced treatment options including durable mechanical circulatory support or heart transplant.

Shared cardiogenic shock definition:

1. Systolic blood pressure < 90 mmHg for > 30 minutes or need for vasopressors use to maintain systolic blood pressure > 90 mmHg
2. Lactate level > 2.0 mmol/L
3. Pulmonary capillary wedge pressure or left ventricle end diastolic pressure > 15 mmHg (excluding pulmonary embolism)
4. Cardiac Index ≤ 2.2 l/min/m2
5. Diuresis < 30 ml/h
6. Clinical signs of peripheral hypoperfusion

Data required by "hub" from "spoke"

1. Echocardiography with data on left and right ventricle function
2. Current aortic and mixed venous blood gases
3. Pulmonary artery catheter measurements including calculation of cardiac power, pulmonary artery pulsatile index, cardiac output, cardiac index, pulmonary artery wedge pressure, pulmonary vascular resistance, systemic vascular resistance (excluding pulmonary embolism)
4. Peripheral blood tests including liver and kidney function, morphology, troponin, natriuretic peptides
5. Currently used and possible for use vascular accesses
6. For pulmonary embolism: computed tomography of pulmonary arteries

Upon telephone contact "hub" shock team decides on patients transfer or further treatment in "spoke" facility. When decision on transfer is taken shock team members gather at emergency room when patient arrives and decides on treatment options according to shock team protocol. As a "hub" Wroclaw University Hospital provides mechanical circulatory support (Intra-aortic balloon pump, Impella CP (Cardiac Power), Impella 5.0, Impella RP (Right Pump), ECMO (ExtraCorporeal Membrane Oxygenation), Levitronix, HeartMate3) together with heart transplant program as a regional reference center for advanced heart failure patients. Additionally for acute pulmonary embolism complicated by shock "hub" provides peripheral or local thrombolysis and in case of contraindication for thrombolysis - transcatheter thrombectomy or surgical embolectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilled definition of cardiogenic shock
2. Age 18 - 60 years
3. Shock duration below 24 hours

Exclusion Criteria:

1. History of cardiac arrest with anoxemic brain injury
2. Irreversible multiorgan failure
3. End stage of chronic diseases other than heart failure
4. Neoplastic disease
5. Lack of vascular access

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: LSCSI is designed to treat cardiogenic shock which may develop during:
  1. Acute coronary syndrome
  2. Acute decompensated heart failure
  3. Acute myocarditis
  4. Acute or decompensated chronic valvular heart disease
  5. Takotsubo cardiomyopathy
  6. Peripartum cardiomyopathy
  7. Acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
30-days all-cause mortality | 30 days
  All-cause mortality

SECONDARY OUTCOMES:
12-months mortality | 12 months
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Heart Disease of Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided